CLINICAL TRIAL: NCT02742935
Title: A Phase 1 Clinical Study on the Safety and Tolerability of PD-1 Antibody SHR-1210 in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety and Tolerability of Using SHR-1210 by Advanced Solid Tumor Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-103
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor; Breast Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- camrelizumab (Experimental): camrelizumab (SHR-1210) injection, 60,200,400mg/dose, intravenous infusion over 30 minutes, every 2 weeks.
  Interventions: Biological: camrelizumab

INTERVENTIONS:
Biological: camrelizumab — A fully humanized anti-PD-1 monoclonal immunoglobulin (IgG4 subtype)
  Other Names: SHR-1210

SUMMARY:
This is an open-label, non-randomized, dose escalation phase I trial to evaluate safety and tolerability of SHR-1210 in patients with advanced solid tumors. The primary objective is to assess safety and tolerability of SHR-1210 and identify recommended phase II doses of SHR-1210 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, nonrandomized, dose-escalation Phase 1 study to evaluate safety and tolerability of SHR-1210 in subjects with advanced Solid Tumors who have failed current standard antitumor therapies.

The safety and tolerability of SHR-1210 will be assessed by ongoing reviews of clinical laboratory tests, Eastern Cooperative Oncology Group (ECOG) performance status, physical examination, electrocardiogram (ECG), and adverse events. Evaluations of immune safety will also be conducted (immune-related AEs, or labs of autoimmune sera, inflammatory events, and immunogenicity). Safety evaluations (both clinical and laboratory) are performed at baseline, before each study treatment, and throughout the study.

Efficacy will be assessed every 8 weeks. The study consists of 3 periods: screening (up to 14 days before the first dose), treatment, and follow-up (up to 90 days after the last dose of study treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-65 years of age;
2. Histologically confirmed solid tumor ;
3. Documented as advanced disease(unresectable or metastatic disease), failure to standard therapies or lack of standard therapy;
4. ECOG performance status of 0 or 1;
5. Life expectancy ≥ 12 weeks.;
6. Ideally, subjects enrolled have measurable lesion(s) according to RECIST v1.1/mRECIST(liver cancer);
7. Adequate laboratory parameters during the screening period as evidenced by the following:

   1. Absolute neutrophil count ≥ 1.5 × 109/L ;
   2. Platelets ≥ 100 × 109/L;
   3. Hemoglobin ≥ 9.0 g/dL;
   4. Albumin (ALB) levels ≥ 2.8 g/dL
   5. Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), ALT and AST ≤ 1.5

      * ULN; for subjects with liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN;
   6. Creatinine clearance≥50 mL/min;
8. Female and male who have reproductive potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 3 months after receiving the last dose of study treatment. Women of childbearing potential with pregnancy test negative within 7days before entering the group and not in in lactation;
9. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Subjects with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy, asthma that requires intermittent use of bronchodilators can not be included;
2. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before entering the group;

3 History of organ transplantation (except corneal transplantation);

4. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR-1210 formulation;

5 History or concurrent with other malignant disease, except completely cured basal cell skin cancers and carcinoma in situs of cervix;

6. Presence of symptomatic central nervous system (CNS) metastases (indicated cerebral edema, steroid requirement, or progressive disease), Subjects with brain or meningeal metastases that were previously treated must be clinically stable (MRI) for at least 2 months, and have discontinued systemic steroids (> 10 mg/day prednisone or equivalent) for at least 2 weeks before study drug administration;

7. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) >2 NYHA 2 congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;

8. Prior radiotherapy, systemic chemotherapy (< 6 weeks if chemotherapy including nitrosoureas or mitomycin), hormone therapy, surgery or target therapy within 4 weeks before the study drug administration, or any unresolved AEs > CTC-AE Grade 1;

9. Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);

10. History of immunodeficiency (HIV) or active hepatitis;

11. Participation in a clinical study or less than 1 month from the last dose of investigational drug to sign ICF;

12. May require for other systemic anti-tumor therapy during the study period;

13. History of PD-1/PD-L1 therapy;

14. History of psychotropic substance abuse, alcoholism or drug abuse;

15. Other factors that may lead to the termination of the participation in the study at the discretion of the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
The severity of adverse events (AEs) determined as per NCI CTCAE V4.03. | 28 days
  safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Qing Yang, Doctor, Study Director — Jiangsu Hengrui Pharmaceutical Co., Ltd.
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided